CLINICAL TRIAL: NCT00820690
Title: Gene Expression Signature and Immunohistochemical Markers Associated With Response to Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer
Acronym: LABC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: 135/2008
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
Keywords: neoadjuvant chemotherapy; advanced breast cancer; microarray; correlation analysis; oncoplastic surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; X-Rays; Surgical Procedures, Operative; Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen tissue; parafin tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinical stage III: Women with invasive breast cancer; clinical stage III, condition to receive neoadjuvant chemotherapy based in doxorubicin/ cyclophosphamide and paclitaxel followed by surgery (mastectomy and axillary lymph node dissection)
  Interventions: Drug: doxorubicin; Drug: cyclophosphamide; Drug: paclitaxel; Procedure: Surgery

INTERVENTIONS:
Drug: doxorubicin — 4 cycles AC: doxorubicin 60mg/m2
  Other Names: clinical and radiologic response
Drug: cyclophosphamide — 4 cycles AC: cyclophosphamide 600mg/m2
  Other Names: clinical and radiologic response
Drug: paclitaxel — 4 cycles T: paclitaxel 175mg/m2 after 4 AC
  Other Names: clinical, radiologic and pathologic response
Procedure: Surgery — The surgery will be performed 30 days after the chemotherapy. The correlation between clinical, radiologic and pathologic response will be reported.
  The oncoplastic surgery rate will be reported
  Other Names: Oncoplastic surgery; Mastectomy

SUMMARY:
The purpose of this study is to analyze gene expression signature and immunohistochemical markers associated with clinical and pathological response to neoadjuvant chemotherapy in locally advanced breast cancer.

DETAILED DESCRIPTION:
Locally advanced breast cancer is a common condition in development countries. Neoadjuvant chemotherapy gives the opportunity to identify genetic signatures associated with objective clinical and pathological complete responses.

Patients will receive doxorubicin/cyclophosphamide with paclitaxel. Tumor samples collected before and after chemotherapy will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women with locally advanced women breast cancer
* Histology: ductal ou lobular invasive histology
* Agreement to take part in the study and signature of the informed consent
* Clinical condition to receive doxorubicin/cyclophosphamide and paclitaxel
* ECOG 0 or I

Exclusion Criteria:

* Not clinical stage III
* Inflammatory breast cancer
* Previous treatment
* Previous diagnosis of cancer (except basal cell or squamous cell skin carcinoma and non-invasive cervical carcinoma)
* Pregnancy
* Absence of clinical condition to receive chemotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women breast cancer, clinical stage III; condition to chemotherapy with doxorubicin/cyclophosphamide and paclitaxel
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2012-04 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Clinical objective and pathological responses to chemotherapy | 8 months
  Clinical and radiological examinations to be performed before chemotherapy, after the 4 cycle of AC and before surgery.
  Pathologic evaluation to be performed 30 days after the last cycle of chemotherapy, i.g. after surgery.

SECONDARY OUTCOMES:
Clinical, radiologic and pathologic correlation | 3 years
  tumor concordance measurement among pre-operative physical examination (PE), mammography (MG), ultrasound (US), breast MRI and post-operative pathologic measurement concordance with PE, MG, US and MRI
Surgery | 5 years
  The use and security of oncoplastic surgery after neoadjuvant chemotherapy
Overall actuarial survival | 5 years
Pathologic complete response | 9 months
  Pathologic complete response after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Maria Aparecida A Koike Folgueira, MD, PhD, Study Chair — Faculdade de Medicina - Universidade de São Paulo
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

REFERENCES:
- [Background] Folgueira MA, Carraro DM, Brentani H, Patrao DF, Barbosa EM, Netto MM, Caldeira JR, Katayama ML, Soares FA, Oliveira CT, Reis LF, Kaiano JH, Camargo LP, Vencio RZ, Snitcovsky IM, Makdissi FB, e Silva PJ, Goes JC, Brentani MM. Gene expression profile associated with response to doxorubicin-based therapy in breast cancer. Clin Cancer Res. 2005 Oct 15;11(20):7434-43. doi: 10.1158/1078-0432.CCR-04-0548. PMID 16243817
- [Background] Andre F, Mazouni C, Hortobagyi GN, Pusztai L. DNA arrays as predictors of efficacy of adjuvant/neoadjuvant chemotherapy in breast cancer patients: current data and issues on study design. Biochim Biophys Acta. 2006 Dec;1766(2):197-204. doi: 10.1016/j.bbcan.2006.08.002. Epub 2006 Aug 9. PMID 16962247
- [Background] Apple SK, Suthar F. How do we measure a residual tumor size in histopathology (the gold standard) after neoadjuvant chemotherapy? Breast. 2006 Jun;15(3):370-6. doi: 10.1016/j.breast.2005.08.002. Epub 2005 Sep 26. PMID 16185870
- [Background] Carey LA, Dees EC, Sawyer L, Gatti L, Moore DT, Collichio F, Ollila DW, Sartor CI, Graham ML, Perou CM. The triple negative paradox: primary tumor chemosensitivity of breast cancer subtypes. Clin Cancer Res. 2007 Apr 15;13(8):2329-34. doi: 10.1158/1078-0432.CCR-06-1109. PMID 17438091
- [Background] Eltahir A, Heys SD, Hutcheon AW, Sarkar TK, Smith I, Walker LG, Ah-See AK, Eremin O. Treatment of large and locally advanced breast cancers using neoadjuvant chemotherapy. Am J Surg. 1998 Feb;175(2):127-32. doi: 10.1016/s0002-9610(97)00279-1. PMID 9515529
- [Background] Fernandez-Sanchez M, Gamboa-Dominguez A, Uribe N, Garcia-Ulloa AC, Flores-Estrada D, Candelaria M, Arrieta O. Clinical and pathological predictors of the response to neoadjuvant anthracycline chemotherapy in locally advanced breast cancer. Med Oncol. 2006;23(2):171-83. doi: 10.1385/MO:23:2:171. PMID 16720917
- [Background] Mamounas EP, Bryant J, Lembersky B, Fehrenbacher L, Sedlacek SM, Fisher B, Wickerham DL, Yothers G, Soran A, Wolmark N. Paclitaxel after doxorubicin plus cyclophosphamide as adjuvant chemotherapy for node-positive breast cancer: results from NSABP B-28. J Clin Oncol. 2005 Jun 1;23(16):3686-96. doi: 10.1200/JCO.2005.10.517. Epub 2005 May 16. PMID 15897552
- [Background] Fisher B, Bryant J, Wolmark N, Mamounas E, Brown A, Fisher ER, Wickerham DL, Begovic M, DeCillis A, Robidoux A, Margolese RG, Cruz AB Jr, Hoehn JL, Lees AW, Dimitrov NV, Bear HD. Effect of preoperative chemotherapy on the outcome of women with operable breast cancer. J Clin Oncol. 1998 Aug;16(8):2672-85. doi: 10.1200/JCO.1998.16.8.2672. PMID 9704717
- [Background] Goldstein NS, Decker D, Severson D, Schell S, Vicini F, Margolis J, Dekhne NS. Molecular classification system identifies invasive breast carcinoma patients who are most likely and those who are least likely to achieve a complete pathologic response after neoadjuvant chemotherapy. Cancer. 2007 Oct 15;110(8):1687-96. doi: 10.1002/cncr.22981. PMID 17722109
- [Background] Keam B, Im SA, Kim HJ, Oh DY, Kim JH, Lee SH, Chie EK, Han W, Kim DW, Moon WK, Kim TY, Park IA, Noh DY, Heo DS, Ha SW, Bang YJ. Prognostic impact of clinicopathologic parameters in stage II/III breast cancer treated with neoadjuvant docetaxel and doxorubicin chemotherapy: paradoxical features of the triple negative breast cancer. BMC Cancer. 2007 Nov 1;7:203. doi: 10.1186/1471-2407-7-203. PMID 17976237
- [Background] Kuerer HM, Newman LA, Smith TL, Ames FC, Hunt KK, Dhingra K, Theriault RL, Singh G, Binkley SM, Sneige N, Buchholz TA, Ross MI, McNeese MD, Buzdar AU, Hortobagyi GN, Singletary SE. Clinical course of breast cancer patients with complete pathologic primary tumor and axillary lymph node response to doxorubicin-based neoadjuvant chemotherapy. J Clin Oncol. 1999 Feb;17(2):460-9. doi: 10.1200/JCO.1999.17.2.460. PMID 10080586
- [Background] Kurosumi M. Significance and problems in evaluations of pathological responses to neoadjuvant therapy for breast cancer. Breast Cancer. 2006;13(3):254-259. doi: 10.2325/jbcs.13.254. PMID 16929118
- [Background] Molina R, Filella X, Zanon G, Pahisa J, Alicarte J, Munoz M, Farrus B, Ballesta AM. Prospective evaluation of tumor markers (c-erbB-2 oncoprotein, CEA and CA 15.3) in patients with locoregional breast cancer. Anticancer Res. 2003 Mar-Apr;23(2A):1043-50. PMID 12820345
- [Background] Prisack HB, Karreman C, Modlich O, Audretsch W, Danae M, Rezai M, Bojar H. Predictive biological markers for response of invasive breast cancer to anthracycline/cyclophosphamide-based primary (radio-)chemotherapy. Anticancer Res. 2005 Nov-Dec;25(6C):4615-21. PMID 16334152
- [Background] Rouzier R, Mathieu MC, Sideris L, Youmsi E, Rajan R, Garbay JR, Andre F, Marsiglia H, Spielmann M, Delaloge S. Breast-conserving surgery after neoadjuvant anthracycline-based chemotherapy for large breast tumors. Cancer. 2004 Sep 1;101(5):918-25. doi: 10.1002/cncr.20491. PMID 15329898
- [Background] Schott AF, Roubidoux MA, Helvie MA, Hayes DF, Kleer CG, Newman LA, Pierce LJ, Griffith KA, Murray S, Hunt KA, Paramagul C, Baker LH. Clinical and radiologic assessments to predict breast cancer pathologic complete response to neoadjuvant chemotherapy. Breast Cancer Res Treat. 2005 Aug;92(3):231-8. doi: 10.1007/s10549-005-2510-1. PMID 16155794
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] van der Hage JA, van de Velde CJ, Julien JP, Tubiana-Hulin M, Vandervelden C, Duchateau L. Preoperative chemotherapy in primary operable breast cancer: results from the European Organization for Research and Treatment of Cancer trial 10902. J Clin Oncol. 2001 Nov 15;19(22):4224-37. doi: 10.1200/JCO.2001.19.22.4224. PMID 11709566
- [Background] van der Hage JA, van de Velde CJ, Julien JP, Floiras JL, Delozier T, Vandervelden C, Duchateau L. Improved survival after one course of perioperative chemotherapy in early breast cancer patients. long-term results from the European Organization for Research and Treatment of Cancer (EORTC) Trial 10854. Eur J Cancer. 2001 Nov;37(17):2184-93. doi: 10.1016/s0959-8049(01)00294-5. PMID 11677105
- [Background] Faneyte IF, Schrama JG, Peterse JL, Remijnse PL, Rodenhuis S, van de Vijver MJ. Breast cancer response to neoadjuvant chemotherapy: predictive markers and relation with outcome. Br J Cancer. 2003 Feb 10;88(3):406-12. doi: 10.1038/sj.bjc.6600749. PMID 12569384
- [Derived] Zucca Matthes AG, Uemura G, Kerr L, Matthes AC, Michelli RA, Folgueira MA, da Costa Viera RA. Feasibility of oncoplastic techniques in the surgical management of locally advanced breast cancer. Int J Surg. 2012;10(9):500-5. doi: 10.1016/j.ijsu.2012.07.009. Epub 2012 Jul 31. PMID 22858800